CLINICAL TRIAL: NCT04033445
Title: A Phase 2b/3, Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Protocol to Evaluate the Efficacy and Safety of Guselkumab in Participants With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Study of Guselkumab in Participants With Moderately to Severely Active Ulcerative Colitis
Acronym: QUASAR
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108657; CNTO1959UCO3001 (Other: Janssen Research & Development, LLC); 2018-004002-25 (EudraCT Number); 2023-504718-31-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2019-07-24; First posted 2019-07-26 (Actual); Results first posted 2024-11-18 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — guselkumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Induction Study 1: Guselkumab Dose 1 (Experimental): Participants will receive guselkumab dose 1 intravenously (IV) in Induction Study 1. Subsequent study treatment will be determined by the participant's clinical response status at Week 12.
  Interventions: Drug: Guselkumab
- Induction Study 1: Guselkumab Dose 2 (Experimental): Participants will receive guselkumab dose 2 IV in Induction Study 1. Subsequent study treatment will be determined by the participant's clinical response status at Week 12.
  Interventions: Drug: Guselkumab
- Induction Study 1: Placebo IV (Placebo Comparator): Participants will receive matching placebo IV in Induction Study 1. Subsequent study treatment will be determined by the participant's clinical response status at Week 12. Clinical nonresponders will be administered guselkumab IV.
  Interventions: Drug: Placebo
- Induction Study 2: Guselkumab IV (Experimental): Participants will receive guselkumab IV in Induction Study 2. Subsequent study treatment will be determined by the participant's clinical response status at Week 12.
  Interventions: Drug: Guselkumab
- Induction Study 2: Placebo IV (Placebo Comparator): Participants will receive matching placebo IV in Induction Study 2. Subsequent study treatment will be determined by the participant's clinical response status at Week 12. Clinical nonresponders will be administered guselkumab IV.
  Interventions: Drug: Placebo
- Maintenance Study: Maintenance Dose Regimen 1 (Experimental): Participants will receive guselkumab maintenance dose regimen 1 subcutaneously (SC) every 4 weeks (q4w).
  Interventions: Drug: Guselkumab
- Maintenance Study: Maintenance Dose Regimen 2 (Experimental): Participants will receive guselkumab maintenance dose regimen 2 SC every 8 weeks (q8w).
  Interventions: Drug: Guselkumab
- Maintenance Study: Placebo SC (Placebo Comparator): Participants will receive matching placebo SC q4w.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Participants will receive matching placebo IV or SC.
  Arms: Induction Study 1: Placebo IV; Induction Study 2: Placebo IV; Maintenance Study: Placebo SC
Drug: Guselkumab — Participants will receive guselkumab IV or SC.
  Arms: Induction Study 1: Guselkumab Dose 1; Induction Study 1: Guselkumab Dose 2; Induction Study 2: Guselkumab IV; Maintenance Study: Maintenance Dose Regimen 1; Maintenance Study: Maintenance Dose Regimen 2

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of guselkumab in participants with moderately to severely active ulcerative colitis (UC).

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of ulcerative colitis (UC)
* Moderately to severely active UC, defined by modified Mayo score
* Demonstrated inadequate response or intolerance to medical therapies specified in the protocol
* Screening laboratory test results within the parameters specified in the protocol

Exclusion Criteria:

* Diagnosis of indeterminate colitis, microscopic colitis, ischemic colitis, or Crohn's disease or clinical findings suggestive of Crohn's disease
* UC limited to the rectum only or to less than (<) 20 centimeter (cm) of the colon
* Presence of a stoma
* Presence or history of a fistula
* Receiving prohibited medications and/or treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1064 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2023-09-19 (Actual); Study Completion 2027-09-29 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (388):
- United States (51):
  - Om Research LLC, Lancaster, California
  - UCLA, Los Angeles, California
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Florida Research Network, LLC, Gainesville, Florida
  - University of Florida Health Jacksonville, Gainesville, Florida
  - Harmony Medical Research Institute, Inc., Hialeah, Florida
  - UF Health Jacksonville Gastroenterology Emerson, Jacksonville, Florida
  - I.H.S. Health. LLC, Kissimmee, Florida
  - Columbus Clinical Services LLC, Miami, Florida
  - Vista Health Research, LLC, Miami, Florida
  - Orlando Health, Orlando, Florida
  - Care Access Research, Orlando, Orlando, Florida
  - Synexus Clinical Research US Inc, Pinellas Park, Florida
  - Univ. of South Florida Med. Group, Tampa, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Morehouse School of Medicine, Atlanta, Georgia
  - The Emory Clinic, Atlanta, Georgia
  - Atlanta Center For Gastroenterology, Decatur, Georgia
  - Gastroenterolgy Associates of Central GA, Macon, Georgia
  - University of Chicago, Chicago, Illinois
  - Health Science Research Center, Pratt, Kansas
  - Tri-State Gastroenterology Assoc, Crestview Hills, Kentucky
  - Baystate Medical Center, Springfield, Massachusetts
  - Clinical Research Institute of Michigan, LLC, Clinton Township, Michigan
  - Revive Research Institute, Farmington Hills, Michigan
  - Infusion Associates, Grand Rapids, Michigan
  - Mid-America Gastro-Intestinal Consultants, Kansas City, Missouri
  - Barnes-jewish Hospital, St Louis, Missouri
  - Las Vegas Medical Research, Las Vegas, Nevada
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Hospital Medical Center, Raleigh, North Carolina
  - Synexus Clinical Research US Inc, Columbus, Ohio
  - Digestive Specialists, Inc, Springboro, Ohio
  - Gastro Intestinal Research Institute of Northern Ohio LLC, Westlake, Ohio
  - Care Access Research, Poland, Youngstown, Ohio
  - Digestive Disease Specialists Inc, Oklahoma City, Oklahoma
  - US Digestive Health, Wyomissing, Pennsylvania
  - Synexus Clinical Research US Inc, Anderson, South Carolina
  - Gastroenterology Associates of Orangeburg, SC, Orangeburg, South Carolina
  - Erlanger Health System, Chattanooga, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Caprock Gastro Research, Lubbock, Texas
  - Tyler Research Institute, LLC, Tyler, Texas
  - Care Access Research, Ogden, Ogden, Utah
  - Care Access Research- Salt Lake City, Salt Lake City, Utah
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
  - UW-Harborview Medical Center, Seattle, Washington
  - Providence Medical Group, Spokane, Washington
  - Velocity Clinical Research Spokane, Spokane, Washington
  - Care Access Research, Casper, Casper, Wyoming
- Argentina (11):
  - CEMIC (Centro de Educación Médica e Investigaciones Clínicas), Buenos Aires
  - Cer Instituto Medico, Buenos Aires
  - CINME Centro de Investigaciones Metabolicas, Buenos Aires
  - Hospital General de Agudos José Maria Ramos Mejía, Buenos Aires
  - Centro Médico Dra. De Salvo, Caba
  - Clinica Adventista Belgrano, Ciudad de Buenos Aires
  - Sanatorio Duarte Quiroz, Córdoba
  - Centro de Investigaciones Medicas Mar Del Plata, Mar del Plata
  - Fundacion de Estudios Clinicos, Rosario
  - Hospital Provincial del Centenario, Rosario
  - Hospital de Alta Complejidad en Red 'El Cruce', San Juan Bautista
- Australia (8):
  - Emeritus Research, Camberwell
  - Monash Health, Clayton
  - Western Health, Footscray
  - Fiona Stanley Hospital, Murdoch
  - Royal Perth Hospital, Perth
  - Mater Hospital, South Brisbane
  - St John of God Subiaco Hospital, Subiaco
  - Princess Alexandra Hospital, Woolloongabba
- Universitaetsklinikum Salzburg Landeskrankenhaus, Salzburg, Austria
- Belgium (7):
  - AZ Sint-Lucas, Bruges
  - CHU Saint-Pierre, Brussels
  - Hopital Erasme, Brussels
  - AZ Maria Middelares, Ghent
  - Universitair Ziekenhuis Gent, Ghent
  - Algemeen Ziekenhuis Jan Palfijn Merksem, Merksem
  - Algemeen Ziekenhuis Delta, Roeselare
- Brazil (14):
  - L2IP Instituto de Pesquisas Clinicas, Brasília
  - Sociedade Campineira de Educacao e Instrucao Hospital e Maternidade Celso Pierro, Campinas
  - CDC - Centro Digestivo de Curitiba, Curitiba
  - Eurolatino Pesquisas Medicas Ltda, Juiz de Fora
  - Instituto Mederi de Pesquisa e Saude, Passo Fundo
  - Hospital das Clinicas de Porto Alegre, Porto Alegre
  - NPCRS Nucleo de Pesquisa Clinica do Rio Grande do Sul, Porto Alegre
  - Universidade Federal do Rio de Janeiro - Faculdade de Medicina, Rio de Janeiro
  - CLIAGEN - Clinica de Atencao em Gastroenterologia Especializada e Nutricao, Salvador
  - CPQuali Pesquisa Clinica LTDA ME, São Paulo
  - BR Trials, São Paulo
  - Onco Star SP Oncologia Ltda, São Paulo
  - Fundacao Universidade Federal do Piaui - Universidade Federal do Piaui, Teresina
  - Eurolatino Pesquisas Medicas Ltda, Uberlândia
- Bulgaria (8):
  - Medical Centre Asklepii OOD, Dupnitsa
  - Medical Center-1-Sevlievo EOOD, Sevlievo
  - 2-nd MHAT, Sofia
  - 4th MHAT - Sofia, Sofia
  - DCC Convex EOOD, Sofia
  - Acibadem City Clinic - Oncology Center, Sofia
  - MHAT 'St. Marina' EAD, Varna
  - MHAT Dr Stefan Cherkezov, Veliko Tarnovo
- Canada (6):
  - G I R I GI Research Institute Foundation, Vancouver, British Columbia
  - Health Sciences Centre, Winnipeg, Manitoba
  - Barrie GI Associates, Barrie, Ontario
  - Toronto Immune and Digestive Health Institute Inc, Toronto, Ontario
  - Hopital Maisonneuve Rosemont, Montreal, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
- China (28):
  - Capital Medical University, Beijing Friendship Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - China-Japan Union Hospital of Jilin University, Changchun
  - The second Xiangya Hospital of Central South University, Changsha
  - The Third Xiangya Hospital of Central Sourth University, Changsha
  - West China Hospital of Sichuan University, Chengdu
  - Daping Hospital, Chongqing
  - The Second Hospital To Dalian Medical University, Dalian
  - First Affiliated Hospital of Gannan Medical University, Ganzhou
  - The First Affiliated Hospital Sun Yat sen University, Guangzhou
  - The Sixth Affiliated Hospital Sun Yat sen University, Guangzhou
  - The First Affiliated Hospital Zhejiang University College of Medicine, Hangzhou
  - The Second Affiliated Hospital of Zhejiang University, Hangzhou
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - First Affiliated Hospital of Kunming Medical Unversity, Kunming
  - The First Affiliated Hospital of NanChang University, Nanchang
  - Nanjing Drum Tower Hospital, Nanjing
  - Zhongda Hospital Southeast University, Nanjing
  - Jiangsu Province Hospital, Nanjing
  - Ruijing Hospital Affiliated To Shanghai Jiaotong University School Of Medicine, Shanghai
  - Shengjing Hospital Of China Medical University, Shenyang
  - The Second Hospital Affiliated To Suzhou University, Suzhou
  - The first affiliated hospital of suzhou University, Suzhou
  - Tianjin Medical University General Hospital, Tianjin
  - Wuhan Union Hospital, Wuhan
  - Tongji Hospital, Tongji Medical College of HUST, Wuhan
  - Wuxi People s Hospital, Wuxi
- Czechia (12):
  - Nemocnice Ceske Budejovice a s, České Budějovice
  - Endohope Havirov s.r.o., Havířov
  - Gastroenterologie, s.r.o., Hradec Kralove, Hradec Kralova
  - MUDr. Gregar s.r.o., Olomouc
  - Vitkovicka nemocnice a.s., Ostrava
  - Artroscan s r o, Ostrava
  - Synexus Czech s.r.o., Prague
  - ResTrial GastroEndo, s.r.o, Prague
  - Nemocnice na Homolce, Prague
  - AXON Clinical s.r.o., Prague
  - ISCARE a.s., Prague
  - Nemocnice Strakonice, a.s., Strakonice
- France (12):
  - CHU caen, Caen
  - Hopital Beaujon, Clichy
  - CHRU de Lille Hopital Claude Huriez, Lille
  - Hopital Saint Eloi, Montpellier
  - CHU de Nice Hopital de l Archet, Nice
  - Hopital Saint Antoine, Paris
  - Hopital Haut-Leveque, CMC Magellan, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU Saint Etienne Hopital Nord, Saint-Priest-en-Jarez
  - Nouvel Hopital Civil, Strasbourg
  - CHU Rangueil, Toulouse
  - CHRU Nancy Brabois, Vandœuvre-lès-Nancy
- Germany (7):
  - Universitaetsklinikum Charite, Campus Virchow Klinikum, Berlin
  - BSF Studiengesellschaft, Halle
  - Medizinische Hochschule Hannover, Hanover
  - Praxisgemeinschaft Jerichow, Jerichow
  - Staedtisches Klinikum Lueneburg, Lüneburg
  - Zentrum für Gastroenterologie Saar MVZ GmbH, Saarbrücken
  - Universitaetsklinikum Ulm, Ulm
- Hungary (8):
  - Synexus Magyarorszag Kft, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Semmelweis University, Budapest
  - Vasutegeszsegugyi Nonprofit Kozhasznu Kft, Debrecen
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Gyongyosi Bugat Pal Korhaz, Gyöngyös
  - Synexus Magyarorszag Kft, Gyula
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Orvostudomanyi Kar, Belgyogyaszati Klinika, Szeged
- Ireland (3):
  - Beaumont Hospital, Dublin
  - St Vincent's University Hospital, Dublin
  - University Hospital Galway - Ireland, Galway
- Israel (7):
  - Rambam Medical Center, Haifa
  - Bnai Zion Medical Center, Haifa
  - Wolfson Medical Center, Holon
  - Shaare Zedek Medical Center, Jerusalem
  - Lev Talpiot Clinic, Jerusalem
  - Galilee Medical Center, Nahariya
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (11):
  - Policlinico Sant'Orsola Malpighi, Bologna
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - Ospedale Classificato Equiparato Sacro Cuore Don Calabria di Negrar, Negrar
  - Azienda Ospedaliera di Padova, Padua
  - Ospedale Villa Sofia-Cervello, Palermo
  - Azienda Ospedaliera G.Salvini Ospedale di Rho, Rho
  - Università Campus Biomedico di Roma, Roma
  - Fondazione Policlinico Gemelli Università Cattolica, Roma
  - Istituto Clinico Humanitas Rozzano, IRCCS, Rozzano
  - Casa Sollievo Della Sofferenza IRCCS, San Giovanni Rotondo
  - AO Ordine Mauriziano, Torino
- Japan (74):
  - Institute of Science Tokyo Hospital, Bunkyō City
  - Juntendo University Hospital Urayasu, Chiba
  - Fukuoka University Chikushi Hospital, Chikushino-shi
  - Ehime Prefectural Central Hospital, Ehime
  - Sai Gastroenterology Proctology, Fujiidera-shi
  - Fukuoka University Hospital, Fukuoka
  - Kitakyushu Municipal Medical Center, Fukuoka-ken
  - Fukushima Medical University Hospital, Fukushima
  - Gifu University Hospital, Gifu
  - Hachinohe City Hospital, Hachinohe
  - Tokai University Hachioji Hospital, Hachiōji
  - Hakodate Goryoukaku Hospital, Hakodate
  - Matsunami General Hospital, Hashima-gun
  - National Hospital Organization Hirosaki General Medical Center, Hirosaki
  - Hirosaki University Hospital, Hirosaki
  - Kure Kyosai Hospital, Hiroshima
  - Asahikawa Medical University Hospital, Hokkaido
  - Mito Saiseikai General Hospital, Ibaraki
  - Shimane University Hospital, Izumo
  - Imamura General Hospital, Kagoshima
  - Kagoshima University Hospital, Kagoshima
  - Izuro Imamura Hospital, Kagoshima
  - Kagoshima IBD Gastroenterology Clinic, Kagoshima
  - Sameshima Hospital, Kagoshima
  - St Marianna University Hospital, Kanagawa
  - Matsushima Hospital, Kanagawa
  - Kanazawa University Hospital, Kanazawa
  - National Hospital Organization Kanazawa Medical Center, Kanazawa
  - Nara Medical University Hospital, Kashihara
  - The Jikei University Kashiwa Hospital, Kashiwa
  - Tsujinaka Hospital Kashiwanoha, Kashiwa
  - Kyushu Rosai Hospital, Kitakyushu
  - Kobe University Hospital, Kobe
  - Aoyama Naika Clinic, Kobe
  - National Hospital Organization Kochi National Hospital, Kochi
  - Yamanashi Prefectural Central Hospital, Kofu
  - Kumagaya General Hospital, Kumagaya-shi
  - National Hospital Organization Kure Medical Center and Chugoku Cancer Center, Kure
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto
  - National Hospital Organization Matsumoto Medical Center, Matsumoto
  - National Hospital Organization Tokyo Medical Center, Meguro Ku
  - Kitasato University Kitasato Institute Hospital, Minatoku
  - Kyorin University Hospital, Mitaka
  - Takagi Clinic, Miyagi
  - Iwate Medical University Uchimaru Medical Center, Morioka
  - Nagoya University Hospital, Nagoya
  - Nagoya City University Hospital, Nagoya
  - Nagaoka Chuo General Hospital, Niigata
  - Hyogo Medical University Hospital, Nishinomiya Shi
  - Nakagami Hospital, Okinawa
  - Japanese Red Cross Osaka Hospital, Osaka
  - Osaka Metropolitan University Hospital, Osaka
  - Izumiotsu Municipal Hospital, Osaka
  - Oita Red Cross Hospital, Ōita
  - Shinbeppu Hospital, Ōita
  - Osaki Citizen Hospital, Ōsaki
  - Japan Community Health Care Organization Saitama Medical Center, Saitama
  - Kindai University Hospital, Sakai
  - Toho University Sakura Medical Center, Sakura
  - Sapporo Tokushukai Hospital, Sapporo
  - Hokkaido P.W.F.A.C. Sapporo-Kosei General Hospital, Sapporo
  - Sapporo Medical University Hospital, Sapporo
  - Sapporo IBD Clinic, Sapporo
  - Sapporo Higashi Tokushukai Hospital, Sapporo
  - Tokyo Yamate Medical Center, Shinjuku-ku
  - Matsuda Hospital, Shizuoka
  - Tokyo Metropolitan Bokutoh Hospital, Sumida Ku
  - Kagawa Prefectural Central Hospital, Takamatsu
  - Tokushima University Hospital, Tokushima
  - The Jikei University Hospital, Tokyo
  - Mie University Hospital, Tsu
  - Yokkaichi Hazu Medical Center, Yokkaichi
  - Yokohama Municipal Citizen's Hospital, Yokohama
  - University of Fukui Hospital, Yoshida
- Jordan (5):
  - Jordan University Hospital, Amman
  - Istishari Hospital, Amman
  - Khalidi Hospital and Medical Center, Amman
  - Irbid Specialty Hospital, Irbid
  - King Abdullah University Hospital, Irbid
- Latvia (3):
  - Pauls Stradins Clinical University Hospital, Riga
  - Health Centre 4 Centre of Diagnostics, Riga
  - Digestive Diseases Centre GASTRO, Riga
- Malaysia (4):
  - Hospital Serdang, Kajang
  - Hospital University Sains Malaysia, Kelantan
  - Pusat Perubatan Universiti Kebangsaan Malaysia, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
- Netherlands (3):
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Radboudumc, Nijmegen
- New Zealand (3):
  - Dunedin Hospital, Dunedin
  - Auckland City Hospital, Grafton
  - Waikato Hospital, Hamilton
- Poland (16):
  - Gastromed Kralisz Romatowski Stachurska Sp. j., Bialystok
  - Centrum Medyczne Medis, Bydgoszcz
  - Centrum Medyczne Plejady, Krakow
  - Centrum Medyczne Promed, Krakow
  - Gastromed ZOZ, Lublin
  - Medicome Sp z o.o., Oświęcim
  - Centrum Medyczne Medyk, Rzeszów
  - Endoskopia Sp z o.o., Sopot
  - Uromed Jakub Koteras Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin
  - GASTROMED Sp. z o.o., Torun
  - Panstwowy Instytut Medyczny Ministerstwa Spraw Wewnetrznych i Administracji, Warsaw
  - Wojskowy Instytut Medyczny, Warsaw
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw
  - Wro Medica, Wroclaw
  - Melita Medical Sp. z o.o., Wroclaw
  - ETG Zamosc, Zamość
- Portugal (5):
  - Centro Hospitalar e Universitário de Coimbra, EPE, Coimbra
  - Uls Santo Antonio - Hosp. Santo Antonio, Porto
  - Uls Sao Joao - Hosp. Sao Joao, Porto
  - Uls de Entre Douro E Vouga - Hosp. Sao Sebastiao, Santa Maria da Feira
  - Centro Hospitalar de Tondela Viseu, EPE, Viseu
- Russia (17):
  - Immanuel Kant Baltic Federal University, Kaliningrad
  - Road Clinical Hospital at the Nizhny Novgorod Station of the Russian Railways, Nizhny Novgorod
  - Medical Center SibNovoMed LLC, Novosibirsk
  - LLC 'Novosibirsk Gastrocentr', Novosibirsk
  - City Clinical Hospital #2, Perm
  - Rostov State Medical University, Rostov-on-Don
  - International Medical Centre SOGAZ, Saint Petersburg
  - All-Russian Center of Emergency and Radiation Medicine MCRS, Saint Petersburg
  - Eco-safety Ltd, Saint Petersburg
  - Medical University Reaviz, Samara
  - NUZ 'Railway Clinical Hospital on Samara station of LLC 'Russian Railways', Samara
  - Saratov Regional Clinical Hospital, Saratov
  - GBUZ Respublican Clinical Hospital n.a. GG Kuvatova, Ufa
  - City Clinical Hospital # 21, Ufa
  - Regional Clinical Hospital, Yaroslavl
  - Medical Center Meditsinskie Tekhnologii, Yekaterinburg
  - OOO MO New Hospital, Yekaterinburg
- Serbia (3):
  - Zvezdara University Medical Center, Belgrade
  - General Hospital 'Dr Radivoj Simonovic', Sombor
  - General Hospital 'Djordje Joanovic', Zrenjanin
- Slovakia (7):
  - FNsP F.D.R. Banska Bystrica, Banská Bystrica
  - Gastroenterology Department GASTROMART s.r.o., Bardejov
  - Gastroenterology Center ASSIDUO, Bratislava
  - Cliniq s.r.o., Bratislava
  - ENDOMED s.r.o, Košice
  - GASTRO I. s.r.o., Prešov
  - Accout Center, s.r.o., Gastroenterologická ambulancia, Šahy
- South Korea (13):
  - Inje University Haeundae Paik Hospital, Busan
  - Yeungnam University Hospital, Daegu
  - Korea University Ansan Hospital, Gyeonggi-do
  - The Catholic university of Korea, St. Vincent's Hospital, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si
  - KyungHee University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Mary s Hospital, Seoul
  - Chung-Ang University Hospital, Seoul
  - Ajou University Hospital, Suwon
- Spain (7):
  - Hosp. Univ. Germans Trias I Pujol, Badalona
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp. Univ. Dr. Josep Trueta, Girona
  - Hosp. Univ. La Paz, Madrid
  - Hosp. Univ. Marques de Valdecilla, Santander
  - Hosp. Virgen Del Rocio, Seville
  - Hosp. Ntra. Sra. de Valme, Seville
- Sweden (2):
  - Karolinska Universitetssjukhuset, Stockholm
  - Uppsala University, Uppsala
- Taiwan (4):
  - Chang-Hua Christian Hospital, Changhua
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Chang-Gung Memorial Hospital, LinKou Branch, Taoyuan District
- Turkey (Türkiye) (12):
  - Hacettepe University Hospital, Ankara
  - Gazi University Hospital, Ankara
  - Trakya University Medical Faculty, Edirne
  - Istanbul University Istanbul Medical Faculty, Istanbul
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Medicana International Istanbul, Istanbul
  - BAU Medical Park Goztepe Hospital, Istanbul
  - Acibadem Kozyatagi Hospital, Istanbul
  - Ege University Medical Faculty, Izmir
  - Dokuz Eylul University Medical Faculty, Izmir
  - Kocaeli University Medical Faculty, Kocaeli
  - Mersin University Medical Faculty Hospital, Mersin
- Ukraine (13):
  - Municipal Non-Profit Enterprise Ivano Frankivsk Regional Clinical Hospital, Ivano-Frankivsk
  - Communal Nonprofit Enterprise 'City Clinical Hospital # 2 N.A. Prof. O.O. Shalimov', Kharkiv
  - SI 'L.T. Maloyi National Institute of Therapy of National Academy of Medical Sciences of Ukraine, Kharkiv
  - Municipal Institution 'Kherson City Clinical Hospital n.a. Y.Y.Karabelesh', Kherson
  - Medical Center 'Ok Clinic' of LLC 'International Institute of Clinical Studies', Kyiv
  - MC PE Sygma, Kyiv
  - Limited Liability Company Progastro Clinic, Lviv
  - Kalyna Center of Modern Medicine, Lviv
  - Municipal Non-profit Enterprise 'Odesa Regional Clinical Hospital' Odesa Regional Council, Odesa
  - Sumy Regional Clinical Hospital a Non-profit Enterprise of Sumy Regional Council, Sumy
  - Municipal institution of Tepnopil Regional Council 'Ternopil University Hospital', Ternopil
  - Health Clinic Limited Liability Company, Vinnytsia
  - Municipal Non-Profit Enterprise M I Pyrohov Vinnytsia Regional Clinical Hospital, Vinnytsia
- United Kingdom (3):
  - Glasgow Royal Infirmary, Glasgow
  - Guy's and St Thomas' Hospital, London
  - St Georges Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Chen B, Ye BD, Cao Q, Hirai F, Saruta M, Chen M, Pelak S, Shipitofsky N, Miao Y, Herr K, Wahking B, Zhuo J, Hisamatsu T. Guselkumab in East Asians With Moderate-to-Severe Ulcerative Colitis: Subgroup Analysis of the QUASAR Induction and Maintenance Studies. J Gastroenterol Hepatol. 2025 Sep;40(9):2197-2208. doi: 10.1111/jgh.17036. Epub 2025 Jun 26. PMID 40574492
- [Derived] Rubin DT, Allegretti JR, Panes J, Shipitofsky N, Yarandi SS, Huang KG, Germinaro M, Wilson R, Zhang H, Johanns J, Feagan BG, Hisamatsu T, Lichtenstein GR, Bressler B, Peyrin-Biroulet L, Sands BE, Dignass A; QUASAR Study Group. Guselkumab in patients with moderately to severely active ulcerative colitis (QUASAR): phase 3 double-blind, randomised, placebo-controlled induction and maintenance studies. Lancet. 2025 Jan 4;405(10472):33-49. doi: 10.1016/S0140-6736(24)01927-5. Epub 2024 Dec 17. PMID 39706209
- [Derived] Peyrin-Biroulet L, Allegretti JR, Rubin DT, Bressler B, Germinaro M, Huang KG, Shipitofsky N, Zhang H, Wilson R, Han C, Feagan BG, Sandborn WJ, Panes J, Hisamatsu T, Lichtenstein GR, Sands BE, Dignass A; QUASAR Study Group. Guselkumab in Patients With Moderately to Severely Active Ulcerative Colitis: QUASAR Phase 2b Induction Study. Gastroenterology. 2023 Dec;165(6):1443-1457. doi: 10.1053/j.gastro.2023.08.038. Epub 2023 Sep 1. PMID 37659673

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study consisted of 3 separate studies: induction study 1 (IS-1), induction study 2 (IS-2) and maintenance study (MS). In IS-1 and IS-2, participants with modified Mayo score (MMS) of 4 to 9 at baseline (Induction Week 0 [Week I-0]) with inadequate response or failed to tolerate conventional or advanced therapy were enrolled.
Pre-assignment Details: IS-1 and IS-2 participants with clinical response (CR) at Week I-12/Week I-24 entered MS. Participants who had no CR at Week I-24 stopped study drug and had safety follow-up up to 12 weeks after last dose. CR: decrease from induction baseline in MMS by greater than or equal to (>=)30 percent (%) and >=2 points, with either >=1 point decrease from baseline in rectal bleeding (RB) subscore/RB subscore of 0 or 1. MMS contained 3 subscores: stool frequency, rectal bleeding and endoscopic subscore.
Groups:
- IS-1: Period 1: Placebo IV at Weeks I-0, I-4 and I-8: Participants received single dose of placebo (matching to guselkumab) intravenous (IV) infusion at Weeks I-0, I-4 and I-8. At Week I-12, participants were evaluated for clinical response. Participants who achieved clinical response at Week I-12 entered the maintenance study and participants who did not achieve clinical response at Week I-12 entered IS-1 Period 2.
- IS-1: Period 1: Guselkumab 200 mg IV at Weeks I-0, I-4 and I-8: Participants received single dose of guselkumab 200 milligrams (mg) IV infusion at Weeks I-0, I-4 and I-8. At Week I-12, participants were evaluated for clinical response. Participants who achieved clinical response at Week I-12 entered the maintenance study and participants who did not achieve clinical response at Week I-12 entered IS-1 Period 2.
- IS-1: Period 1: Guselkumab 400 mg IV at Weeks I-0, I-4 and I-8: Participants received single dose of guselkumab 400 mg IV infusion at Weeks I-0, I-4 and I-8. At Week I-12, participants were evaluated for clinical response. Participants who achieved clinical response at Week I-12 entered the maintenance study and participants who did not achieve clinical response at Week I-12 entered IS-1 Period 2.
- IS-1: Period 2: Guselkumab 200 mg IV at Weeks I-12, I-16 and I-20: Participants who initially received placebo and did not achieve clinical response at IS-1 Period 1 Week I-12 were crossed over to guselkumab and received single dose of guselkumab 200 mg IV infusion and placebo (matching to guselkumab) subcutaneous (SC) injection at Weeks I-12, I-16 and I-20. At Week I-24, participants were re-evaluated for clinical response. Participants who achieved clinical response at Week I-24 entered the maintenance study. Participants who did not achieve clinical response at Week I-24 received no further study drug and had a safety follow-up up to 12 weeks after their last dose of study drug.
- IS-1: Period 2: Guselkumab 200 mg SC at Weeks I-12, I-16 and I-20: Participants who initially received guselkumab 200 mg or 400 mg IV infusion and did not achieve clinical response at IS-1 Period 1 Week I-12 received single dose of guselkumab 200 mg SC injection and placebo (matching to guselkumab) IV infusion at Weeks I-12, I-16 and I-20. At Week I-24, participants were re-evaluated for clinical response. Participants who achieved clinical response at Week I-24 entered the maintenance study. Participants who did not achieve clinical response at Week I-24 received no further study drug and had a safety follow-up up to 12 weeks after their last dose of study drug.
- IS-2: Period 1: Placebo IV at Weeks I-0, I-4 and I-8: Participants received single dose of placebo (matched to guselkumab) IV infusion at Weeks I-0, I-4 and I-8. At Week I-12, participants were evaluated for clinical response. Participants who achieved clinical response at Week I-12 entered the maintenance study. Participants who did not achieve clinical response at Week I-12 entered IS-2 Period 2.
- IS-2: Period 1: Guselkumab 200 mg IV at Weeks I-0, I-4 and I-8: Participants received single dose of guselkumab 200 mg IV infusion at Weeks I-0, I-4 and I-8. At Week I-12, participants were evaluated for clinical response. Participants who achieved clinical response at Week I-12 entered the maintenance study. Participants who did not achieve clinical response at Week I-12 entered IS-2 Period 2.
- IS-2: Period 2: Guselkumab 200 mg IV at Weeks I-12, I-16 and I-20: Participants who initially received placebo and did not achieve clinical response at Week I-12 were crossed over to guselkumab and received guselkumab 200 mg IV infusion and placebo (matching to guselkumab) SC injection at Weeks I-12, I-16 and I-20. At Week I-24, participants were re-evaluated for clinical response. Participants who achieved clinical response at Week I-24 entered the maintenance study. Participants who did not achieve clinical response at Week I-24 received no further study drug and had a safety follow-up up to 12 weeks after their last dose of study drug.
- IS-2: Period 2: Guselkumab 200 mg SC at Weeks I-12, I-16 and I-20: Participants who initially received guselkumab 200 mg IV infusion and did not achieve clinical response at Week I-12 received guselkumab 200 mg SC injection and placebo (matching to guselkumab) IV infusion at Weeks I-12, I-16 and I-20. At Week I-24, participants were re-evaluated for clinical response. Participants who achieved clinical response at Week I-24 entered the maintenance study. Participants who did not achieve clinical response at Week I-24 received no further study drug and had a safety follow-up up to 12 weeks after their last dose of study drug.
- MS: Randomized: Placebo SC Every 4 Weeks (q4w): Participants who achieved clinical response at IS-1 or IS-2 Week I-12 (Period 1) (previously treated with guselkumab) or at Week I-24 (Period 2) (previously treated with placebo and crossover to guselkumab at Week I-12) were randomized to receive placebo (matching to guselkumab) SC injection every 4 weeks (q4w) starting from Week M-0 till Week M-40. Participants who met criteria for loss of clinical response ( that is [i.e.], no longer satisfied the definition of clinical response) underwent single blinded dose adjustment (between Weeks M-8 and M-32) and received guselkumab 200 mg SC injection q4w from the time of dose adjustment through maintenance Week 40.
- MS: Randomized: Guselkumab 100 mg SC q8w: Participants who achieved clinical response at IS-1 or IS-2 Week I-12 (Period 1) (previously treated with guselkumab) or at Week I-24 (Period 2) (previously treated with placebo and crossover to guselkumab at Week I-12) were randomized to receive guselkumab 100 mg SC injection q8w starting from Week M-4 till Week M-36. Participants who met criteria for loss of clinical response (i.e., no longer satisfied the definition of clinical response) underwent single blinded dose adjustment (between Weeks M-8 and M-32) and received guselkumab 200 mg SC injection q4w from the time of dose adjustment through maintenance Week 40.
- MS: Randomized: Guselkumab 200 mg SC q4w: Participants who achieved clinical response at IS-1or IS-2 Week I-12 (Period 1)(previously treated with guselkumab) or at Week I-24 (Period 2) (previously treated with placebo and crossover to guselkumab at Week I-12) were randomized to receive guselkumab 200 mg SC injection q4w starting from Week M-0 till Week M-40. Participants who met criteria for loss of clinical response (i.e., no longer satisfied the definition of clinical response) underwent single blinded dose adjustment (between Weeks M-8 and M-32) and received guselkumab 200 mg SC injection q4w (sham dose adjustment) from the time of dose adjustment through maintenance Week 40.
- MS: Nonrandomized: Placebo SC q4w: Participants who were treated previously with placebo (matched to guselkumab) and achieved clinical response at IS-1 or IS-2 Week I-12 (Period 1) entered in MS and received placebo (matched to guselkumab) SC injection q4w starting from Week M-0 till Week M-40.
- MS: Nonrandomized: Guselkumab 200 mg SC q4w: Participants who were randomized to guselkumab and did not achieve clinical response at IS-1 or IS-2 Week I-12 (period 1) but achieved clinical response at IS-1 or IS-2 Week I-24 (Period 2) entered in MS and received guselkumab 200 mg SC injection q4w starting from Week M-0 till Week M-40.
Period: IS-1 and IS-2 Period 1 (Week 0 to 12)
Arm/Group | IS-1: Period 1: Placebo IV at Weeks I-0, I-4 and I-8 | IS-1: Period 1: Guselkumab 200 mg IV at Weeks I-0, I-4 and I-8 | IS-1: Period 1: Guselkumab 400 mg IV at Weeks I-0, I-4 and I-8 | IS-1: Period 2: Guselkumab 200 mg IV at Weeks I-12, I-16 and I-20 | IS-1: Period 2: Guselkumab 200 mg SC at Weeks I-12, I-16 and I-20 | IS-2: Period 1: Placebo IV at Weeks I-0, I-4 and I-8 | IS-2: Period 1: Guselkumab 200 mg IV at Weeks I-0, I-4 and I-8 | IS-2: Period 2: Guselkumab 200 mg IV at Weeks I-12, I-16 and I-20 | IS-2: Period 2: Guselkumab 200 mg SC at Weeks I-12, I-16 and I-20 | MS: Randomized: Placebo SC Every 4 Weeks (q4w) | MS: Randomized: Guselkumab 100 mg SC q8w | MS: Randomized: Guselkumab 200 mg SC q4w | MS: Nonrandomized: Placebo SC q4w | MS: Nonrandomized: Guselkumab 200 mg SC q4w
Started | 109 | 108 | 111 | 0 | 0 | 296 | 440 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Treated | 108 | 108 | 111 | 0 | 0 | 295 | 440 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Full Analysis Set (FAS) (All randomized participants (in IS-1 and IS-2) with a modified Mayo score (MMS) of 5 to 9 who received at least 1 (partial or complete) dose of study intervention.) | 105 | 101 | 107 | 0 | 0 | 280 | 421 | 0 | 0 | 0 | 0 | 0 | 0 | 0
FAS Participants Who Enrolled Into MS (FAS participants with clinical response status at Week I-12 as determined by the interactive web response system based on the local endoscopy subscore, as prespecified in the protocol.) | 32 | 60 | 65 | 0 | 0 | 82 | 274 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 103 | 105 | 110 | 0 | 0 | 270 | 422 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 3 | 1 | 0 | 0 | 26 | 18 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 1 | 0 | 0 | 0 | 9 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 0 | 0 | 12 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Randomized but not treated | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: IS-1 and IS-2 Period 2 (Week 12 to 24)
Arm/Group | IS-1: Period 1: Placebo IV at Weeks I-0, I-4 and I-8 | IS-1: Period 1: Guselkumab 200 mg IV at Weeks I-0, I-4 and I-8 | IS-1: Period 1: Guselkumab 400 mg IV at Weeks I-0, I-4 and I-8 | IS-1: Period 2: Guselkumab 200 mg IV at Weeks I-12, I-16 and I-20 | IS-1: Period 2: Guselkumab 200 mg SC at Weeks I-12, I-16 and I-20 | IS-2: Period 1: Placebo IV at Weeks I-0, I-4 and I-8 | IS-2: Period 1: Guselkumab 200 mg IV at Weeks I-0, I-4 and I-8 | IS-2: Period 2: Guselkumab 200 mg IV at Weeks I-12, I-16 and I-20 | IS-2: Period 2: Guselkumab 200 mg SC at Weeks I-12, I-16 and I-20 | MS: Randomized: Placebo SC Every 4 Weeks (q4w) | MS: Randomized: Guselkumab 100 mg SC q8w | MS: Randomized: Guselkumab 200 mg SC q4w | MS: Nonrandomized: Placebo SC q4w | MS: Nonrandomized: Guselkumab 200 mg SC q4w
Started | 0 | 0 | 0 | 67 | 79 | 0 | 0 | 172 | 129 | 0 | 0 | 0 | 0 | 0
IS-1: Period 1 Guselkumab 200 mg IV Non Responders | 0 | 0 | 0 | 0 | 38 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
IS-1: Period 1 Guselkumab 400 mg IV Non Responders | 0 | 0 | 0 | 0 | 41 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Treated | 0 | 0 | 0 | 67 | 79 | 0 | 0 | 171 | 129 | 0 | 0 | 0 | 0 | 0
FAS Participants Who Enrolled Into MS (FAS participants with clinical response status at Week I-24 as determined by the interactive web response system based on the local endoscopy subscore, as prespecified in the protocol.) | 0 | 0 | 0 | 49 | 49 | 0 | 0 | 120 | 74 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 64 | 77 | 0 | 0 | 162 | 117 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 10 | 12 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 4 | 6 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Crossed over but not treated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Maintenance Study (Week 0 to Week 44)
Arm/Group | IS-1: Period 1: Placebo IV at Weeks I-0, I-4 and I-8 | IS-1: Period 1: Guselkumab 200 mg IV at Weeks I-0, I-4 and I-8 | IS-1: Period 1: Guselkumab 400 mg IV at Weeks I-0, I-4 and I-8 | IS-1: Period 2: Guselkumab 200 mg IV at Weeks I-12, I-16 and I-20 | IS-1: Period 2: Guselkumab 200 mg SC at Weeks I-12, I-16 and I-20 | IS-2: Period 1: Placebo IV at Weeks I-0, I-4 and I-8 | IS-2: Period 1: Guselkumab 200 mg IV at Weeks I-0, I-4 and I-8 | IS-2: Period 2: Guselkumab 200 mg IV at Weeks I-12, I-16 and I-20 | IS-2: Period 2: Guselkumab 200 mg SC at Weeks I-12, I-16 and I-20 | MS: Randomized: Placebo SC Every 4 Weeks (q4w) | MS: Randomized: Guselkumab 100 mg SC q8w | MS: Randomized: Guselkumab 200 mg SC q4w | MS: Nonrandomized: Placebo SC q4w | MS: Nonrandomized: Guselkumab 200 mg SC q4w
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 201 | 199 | 199 | 122 | 125
Treated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 201 | 199 | 199 | 122 | 125
Full Analysis Set (All participants with a MMS of 5 to 9 who received at least 1 dose (partial or complete) of study intervention in MS, including both randomized and nonrandomized.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 190 | 188 | 190 | 114 | 123
Safety All Randomized and Treated Analysis Set (All participants (regardless of MMS) who were randomized in MS and received at least 1 dose of study intervention in MS.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 203 (2 participants randomized to arm "MS: Randomized: Guselkumab 100 mg SC + Placebo SC" but received placebo only and thus were included in the safety analysis of this arm.) | 197 | 199 | 0 | 0
Dose Adjustment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 75 | 23 | 31 | 0 | 0
Safety All Nonrandomized and Treated Analysis Set (All participants (regardless of MMS) who entered in MS but were not randomized and received at least 1 dose of study intervention in MS.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 122 | 125
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 173 | 177 | 176 | 95 | 107
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 28 | 22 | 23 | 27 | 18
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 9 | 10 | 11 | 5
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 3 | 1 | 5 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 4 | 7 | 6 | 5
Not completed — Non-Compliance With Study Drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 2
Not completed — Site Closure in Ukraine | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) which included all randomized participants (in IS-1 and IS-2) with a modified Mayo score (MMS) of 5 to 9 who received at least 1 (partial or complete) dose of study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | IS-1: Period 1: Placebo IV at Weeks I-0, I-4 and I-8 | IS-1: Period 1: Guselkumab 200 mg IV at Weeks I-0, I-4 and I-8 | IS-1: Period 1: Guselkumab 400 mg IV at Weeks I-0, I-4 and I-8 | IS-2: Period 1: Placebo IV at Weeks I-0, I-4 and I-8 | IS-2: Period 1: Guselkumab 200 mg IV at Weeks I-0, I-4 and I-8 | Total
Number analyzed (Participants) | 105 | 101 | 107 | 280 | 421 | 1014
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.2 (15.05) | 43.3 (14.28) | 40.4 (13.84) | 39.8 (13.43) | 41 (13.9) | 40.9 (13.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 41 | 48 | 119 | 183 | 430
  Male | 66 | 60 | 59 | 161 | 238 | 584
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 4 | 21 | 25 | 59
  Not Hispanic or Latino | 97 | 92 | 98 | 240 | 368 | 895
  Unknown or Not Reported | 4 | 4 | 5 | 19 | 28 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 24 | 23 | 27 | 62 | 88 | 224
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 1
  Black or African American | 1 | 1 | 1 | 3 | 4 | 10
  White | 77 | 73 | 74 | 205 | 304 | 733
  More than one race | 0 | 1 | 0 | 0 | 1 | 2
  Unknown or Not Reported | 3 | 3 | 5 | 10 | 22 | 43
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 0 | 0 | 2 | 5 | 10 | 17
  Australia | 2 | 1 | 2 | 7 | 14 | 26
  Belgium | 1 | 0 | 0 | 3 | 3 | 7
  Brazil | 0 | 2 | 0 | 12 | 15 | 29
  Bulgaria | 1 | 0 | 1 | 2 | 3 | 7
  Canada | 0 | 0 | 0 | 2 | 5 | 7
  China | 7 | 2 | 2 | 26 | 35 | 72
  Czech Republic | 1 | 2 | 1 | 11 | 17 | 32
  France | 5 | 10 | 6 | 10 | 30 | 61
  Germany | 3 | 3 | 3 | 11 | 8 | 28
  Hungary | 4 | 5 | 3 | 11 | 17 | 40
  Ireland | 0 | 0 | 0 | 1 | 0 | 1
  Israel | 0 | 1 | 1 | 5 | 7 | 14
  Italy | 5 | 2 | 6 | 14 | 15 | 42
  Japan | 9 | 12 | 15 | 25 | 33 | 94
  Jordan | 0 | 0 | 0 | 16 | 18 | 34
  Latvia | 0 | 0 | 0 | 5 | 3 | 8
  Malaysia | 0 | 0 | 0 | 3 | 4 | 7
  New Zealand | 0 | 0 | 1 | 2 | 5 | 8
  Poland | 19 | 22 | 24 | 47 | 71 | 183
  Portugal | 2 | 2 | 1 | 1 | 0 | 6
  Russian Federation | 9 | 7 | 6 | 18 | 20 | 60
  Serbia | 0 | 0 | 0 | 5 | 5 | 10
  Slovakia | 0 | 0 | 0 | 2 | 12 | 14
  South Korea | 6 | 7 | 5 | 2 | 11 | 31
  Spain | 2 | 1 | 1 | 2 | 2 | 8
  Sweden | 2 | 1 | 0 | 0 | 3 | 6
  Taiwan | 2 | 1 | 3 | 2 | 1 | 9
  Turkey | 0 | 0 | 2 | 3 | 11 | 16
  Ukraine | 16 | 16 | 14 | 13 | 20 | 79
  United Kingdom | 3 | 1 | 1 | 3 | 6 | 14
  United States | 6 | 3 | 7 | 11 | 17 | 44

OUTCOME MEASURES:

1. Primary Outcome: Induction Study 1: Percentage of Participants With Clinical Response at Week I-12
Description: Clinical response was defined as a decrease from induction baseline in the modified Mayo score by greater than or equal to (>=) 30 percent (%) and >=2 points, with either a >=1 point decrease from baseline (Week 0 of IS-1) in the rectal bleeding subscore or a rectal bleeding subscore of 0 or 1. The modified Mayo scores consisted of 3 subscores: stool frequency, rectal bleeding and endoscopic subscore as determined during central review, each subscore graded from 0 (normal) to 3 (severe) with higher scores indicating more severe disease. These individual subscores were summed up to give a total modified Mayo score range of 0 (normal) to 9 (severe disease), where higher scores indicated more severe disease activity. This outcome measure was planned to be analyzed for specified arms only.
Time Frame: At Week I-12
Population: FAS: all randomized participants (in IS-1) with a modified Mayo score of 5 to 9 who received at least 1 (partial or complete) dose of study intervention.
Measure: Number; unit: Percentage of participants
Arm/Group | IS-1: Period 1: Placebo IV at Weeks I-0, I-4 and I-8 | IS-1: Period 1: Guselkumab 200 mg IV at Weeks I-0, I-4 and I-8 | IS-1: Period 1: Guselkumab 400 mg IV at Weeks I-0, I-4 and I-8
Number analyzed (Participants) | 105 | 101 | 107
Percentage of participants | 27.6 | 61.4 | 60.7
Statistical Analysis 1: Comparison: IS-1: Period 1: Placebo IV at Weeks I-0, I-4 and I-8 vs IS-1: Period 1: Guselkumab 200 mg IV at Weeks I-0, I-4 and I-8; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel (CMH) chi-square; Adjusted treatment difference = 33.6, 95% CI 2-sided [20.9 to 46.3] — Treatment difference between guselkumab group and placebo group was adjusted with CMH weight
Statistical Analysis 2: Comparison: IS-1: Period 1: Placebo IV at Weeks I-0, I-4 and I-8 vs IS-1: Period 1: Guselkumab 400 mg IV at Weeks I-0, I-4 and I-8; Test type: Superiority; p < 0.001, CMH chi-square test; Adjusted treatment difference = 33.1, 95% CI 2-sided [20.8 to 45.4] — Treatment difference between guselkumab group and placebo group was adjusted with CMH weight

2. Primary Outcome: Induction Study 2: Percentage of Participants With Clinical Remission at Week I-12
Description: Clinical remission was based on the modified Mayo score. Clinical remission was defined as Mayo stool frequency subscore of 0 or 1 and not increased from baseline (Week 0 of IS-2), a Mayo rectal bleeding subscore of 0, and Mayo endoscopic subscore of 0 or 1 with no friability. The modified Mayo scores consisted of 3 subscores: stool frequency, rectal bleeding and endoscopic subscore as determined during central review, each subscore graded from 0 (normal) to 3 (severe) with higher scores indicating more severe disease. These individual subscores were summed up to give a total modified Mayo score range of 0 (normal) to 9 (severe disease), where higher scores indicated more severe disease activity. This outcome measure was planned to be analyzed for specified arms only.
Time Frame: At Week I-12
Population: Full analysis set included all randomized participants (in IS-2) with a modified Mayo score of 5 to 9 who received at least 1 (partial or complete) dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | IS-2: Period 1: Placebo IV at Weeks I-0, I-4 and I-8 | IS-2: Period 1: Guselkumab 200 mg IV at Weeks I-0, I-4 and I-8
Number analyzed (Participants) | 280 | 421
Percentage of participants | 7.9 [4.7 to 11.0] | 22.6 [18.6 to 26.6]
Statistical Analysis 1: Comparison: IS-2: Period 1: Placebo IV at Weeks I-0, I-4 and I-8 vs IS-2: Period 1: Guselkumab 200 mg IV at Weeks I-0, I-4 and I-8; Test type: Superiority; p < 0.001, CMH chi-square test; Adjusted treatment difference = 14.9, 95% CI 2-sided [9.9 to 19.9] — Treatment difference between guselkumab group and placebo group was adjusted with CMH weight

3. Primary Outcome: Maintenance Study: Percentage of Participants With Clinical Remission at Week M-44
Description: Clinical remission was based on the modified Mayo score. Clinical remission was defined as Mayo stool frequency subscore of 0 or 1 and not increased from baseline (Week 0 of IS-1 and IS-2), a Mayo rectal bleeding subscore of 0, and Mayo endoscopic subscore of 0 or 1 with no friability. The modified Mayo scores consisted of 3 subscores: stool frequency, rectal bleeding and endoscopic subscore as determined during central review, each subscore graded from 0 (normal) to 3 (severe) with higher scores indicating more severe disease. These individual subscores were summed up to give a total modified Mayo score range of 0 (normal) to 9 (severe disease), where higher scores indicated more severe disease activity. This outcome measure was planned to be analyzed for randomized arms only.
Time Frame: At Week M-44
Population: Randomized full analysis set included all participants with a modified Mayo score of 5 to 9 who were randomized and received at least 1 (partial or complete) dose of study intervention in the maintenance study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MS: Randomized: Placebo SC Every 4 Weeks (q4w) | MS: Randomized: Guselkumab 100 mg SC q8w | MS: Randomized: Guselkumab 200 mg SC q4w
Number analyzed (Participants) | 190 | 188 | 190
Percentage of participants | 18.9 [13.4 to 24.5] | 45.2 [38.1 to 52.3] | 50.0 [42.9 to 57.1]
Statistical Analysis 1: Comparison: MS: Randomized: Placebo SC Every 4 Weeks (q4w) vs MS: Randomized: Guselkumab 100 mg SC q8w; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted treatment difference = 25.2, 95% CI 2-sided [16.4 to 33.9] — Treatment difference between guselkumab group and placebo group was adjusted with CMH weight
Statistical Analysis 2: Comparison: MS: Randomized: Placebo SC Every 4 Weeks (q4w) vs MS: Randomized: Guselkumab 200 mg SC q4w; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted treatment difference = 29.5, 95% CI 2-sided [20.9 to 38.1] — Treatment difference between guselkumab group and placebo group was adjusted with CMH weight

4. Secondary Outcome: Induction Study 1: Percentage of Participants With Clinical Remission at Week I-12
Time Frame: At Week I-12
Reporting Status: Not Posted, anticipated posting 2028-10

5. Secondary Outcome: Induction Study 1: Percentage of Participants With Symptomatic Remission at Week I-12
Time Frame: At Week I-12
Reporting Status: Not Posted, anticipated posting 2028-10

6. Secondary Outcome: Induction Study 1: Percentage of Participants With Endoscopic Healing at Week I-12
Time Frame: At Week I-12
Reporting Status: Not Posted, anticipated posting 2028-10

7. Secondary Outcome: Induction Study 1: Percentage of Participants With Histologic-Endoscopic Mucosal Healing at Week I-12
Time Frame: At Week I-12
Reporting Status: Not Posted, anticipated posting 2028-10

8. Secondary Outcome: Induction Study 1: Percentage of Participants With Endoscopic Normalization at Week I-12
Time Frame: At Week I-12
Reporting Status: Not Posted, anticipated posting 2028-10

9. Secondary Outcome: Induction Study 2: Percentage of Participants With Symptomatic Remission at Week I-12
Time Frame: At Week I-12
Reporting Status: Not Posted, anticipated posting 2028-10

10. Secondary Outcome: Induction Study 2: Percentage of Participants With Endoscopic Healing at Week I-12
Time Frame: At Week I-12
Reporting Status: Not Posted, anticipated posting 2028-10

11. Secondary Outcome: Induction Study 2: Percentage of Participants With Clinical Response at Week I-12
Time Frame: At Week I-12
Reporting Status: Not Posted, anticipated posting 2028-10

12. Secondary Outcome: Induction Study 2: Percentage of Participants With Symptomatic Remission at Week I-4
Time Frame: At Week I-4
Reporting Status: Not Posted, anticipated posting 2028-10

13. Secondary Outcome: Induction Study 2: Percentage of Participants With Inflammatory Bowel Disease Questionnaire (IBDQ) Remission at Week I-12
Time Frame: At Week I-12
Reporting Status: Not Posted, anticipated posting 2028-10

14. Secondary Outcome: Induction Study 2: Percentage of Participants With Histologic-Endoscopic Mucosal Healing at Week I-12
Time Frame: At Week I-12
Reporting Status: Not Posted, anticipated posting 2028-10

15. Secondary Outcome: Induction Study 2: Percentage of Participants With Fatigue Response at Week I-12
Time Frame: At Week I-12
Reporting Status: Not Posted, anticipated posting 2028-10

16. Secondary Outcome: Induction Study 2: Percentage of Participants With Symptomatic Remission at Week I-2
Time Frame: At Week I-2
Reporting Status: Not Posted, anticipated posting 2028-10

17. Secondary Outcome: Induction Study 2: Percentage of Participants With Endoscopic Normalization at Week I-12
Time Frame: At Week I-12
Reporting Status: Not Posted, anticipated posting 2028-10

18. Secondary Outcome: Maintenance Study: Percentage of Participants With Symptomatic Remission at Week M-44
Time Frame: At Week M-44
Reporting Status: Not Posted, anticipated posting 2028-10

19. Secondary Outcome: Maintenance Study: Percentage of Participants With Endoscopic Healing at Week M-44
Time Frame: At Week M-44
Reporting Status: Not Posted, anticipated posting 2028-10

20. Secondary Outcome: Maintenance Study: Percentage of Participants With Corticosteroid-free Clinical Remission at Week M-44
Time Frame: At Week M-44
Reporting Status: Not Posted, anticipated posting 2028-10

21. Secondary Outcome: Maintenance Study: Percentage of Participants With Clinical Response at Week M-44
Time Frame: At Week M-44
Reporting Status: Not Posted, anticipated posting 2028-10

22. Secondary Outcome: Maintenance Study: Percentage of Participants With Histologic-Endoscopic Mucosal Healing at Week M-44
Time Frame: At Week M-44
Reporting Status: Not Posted, anticipated posting 2028-10

23. Secondary Outcome: Maintenance Study: Percentage of Participants With IBDQ Remission at Week M-44
Time Frame: At Week M-44
Reporting Status: Not Posted, anticipated posting 2028-10

24. Secondary Outcome: Maintenance Study: Percentage of Participants With Fatigue Response at Week M-44
Time Frame: At Week M-44
Reporting Status: Not Posted, anticipated posting 2028-10

25. Secondary Outcome: Maintenance Study: Percentage of Participants With Clinical Remission at Week 44 Among the Participants Who Had Achieved Clinical Remission at Maintenance Baseline
Time Frame: At Week M-44
Reporting Status: Not Posted, anticipated posting 2028-10

26. Secondary Outcome: Maintenance Study: Percentage of Participants With Endoscopic Normalization at Week M-44
Time Frame: At Week M-44
Reporting Status: Not Posted, anticipated posting 2028-10

ADVERSE EVENTS:
Time Frame: IS-1 and 2 Period 1: From Week I-0 to Week I-12; IS-1 and 2 Period 2: From Week I-12 to 12 weeks after last dose of study drug (up to 32 weeks); MS: from Week M-0 up to Week M-44
Description: All-cause mortality:Analyzed on all randomized (IS-1 & 2) and enrolled participants (MS). SAEs/Other AEs:IS-1 & 2:All treated analysis set:all randomized participants (regardless of MMS), received at least 1 dose of drug, MS:Safety all randomized and treated analysis set:all participants (regardless of MMS) randomized and received at least 1 dose drug; Safety all nonrandomized and treated analysis set:all non-randomized participants (regardless of MMS) in MS and received at least 1 dose of drug.
Groups:
- MS: Randomized: Placebo SC Every 4 Weeks (q4w): Participants who achieved clinical response at IS-1 or IS-2 Week I-12 (Period 1) (previously treated with guselkumab) or at Week I-24 (Period 2) (previously treated with placebo and crossover to guselkumab at Week I-12) were randomized to receive placebo (matching to guselkumab) SC injection every 4 weeks (q4w) starting from Week M-0 till Week M-40.
- MS: Randomized: Guselkumab 100 mg SC q8w: Participants who achieved clinical response at IS-1 or IS-2 Week I-12 (Period 1) (previously treated with guselkumab) or at Week I-24 (Period 2) (previously treated with placebo and crossover to guselkumab at Week I-12) were randomized to receive guselkumab 100 mg SC injection q8w starting from Week M-4 till Week M-36.
- MS: Randomized: Guselkumab 200 mg SC q4w: Participants who achieved clinical response at IS-1or IS-2 Week I-12 (Period 1)(previously treated with guselkumab) or at Week I-24 (Period 2) (previously treated with placebo and crossover to guselkumab at Week I-12) were randomized to receive guselkumab 200 mg SC injection q4w starting from Week M-0 till Week M-40.
- MS: Dose Adjustment: Placebo SC q4w to Guselkumab 200 mg SC q4w: Participants who achieved clinical response in IS-1 or IS-2 (at Week I-12 or Week I-24) and randomized in MS to receive placebo (matched to guselkumab) SC injection and met criteria for loss of clinical response (i.e., no longer satisfied the definition of clinical response) underwent single blinded dose adjustment (between Weeks M-8 and M-32) and received guselkumab 200 mg SC injection q4w from the time of dose adjustment through maintenance Week 40.
- MS: Dose Adjustment: Guselkumab 100 mg SC q8w to Guselkumab 200 mg SC q4w: Participants who achieved clinical response in IS-1 or IS-2 (at Week I-12 or Week I-24) and randomized in MS to receive guselkumab 100 mg SC injection q4w and met criteria for loss of clinical response (i.e., no longer satisfied the definition of clinical response) underwent single blinded dose adjustment (between Weeks M-8 and M-32) and received guselkumab 200 mg SC injection q4w from the time of dose adjustment through maintenance Week 40.
- MS: Dose Adjustment: Guselkumab 200 mg SC q4w to Guselkumab 200 mg SC q4w: Participants who achieved clinical response in IS-1 or IS-2 (at Week I-12 or Week I-24) and randomized in MS to receive guselkumab 200 mg SC injection q4w and met criteria for loss of clinical response (i.e., no longer satisfied the definition of clinical response) underwent single blinded dose adjustment (between Weeks M-8 and M-32) and received guselkumab 200 mg SC injection q4w (sham dose adjustment) from the time of dose adjustment through maintenance Week 40.
Arm/Group | IS-1: Period 1: Placebo IV at Weeks I-0, I-4 and I-8 | IS-1: Period 1: Guselkumab 200 mg IV at Weeks I-0, I-4 and I-8 | IS-1: Period 1: Guselkumab 400 mg IV at Weeks I-0, I-4 and I-8 | IS-1: Period 2: Guselkumab 200 mg IV at Weeks I-12, I-16 and I-20 | IS-1: Period 2: Guselkumab 200 mg SC at Weeks I-12, I-16 and I-20 | IS-2: Period 1: Placebo IV at Weeks I-0, I-4 and I-8 | IS-2: Period 1: Guselkumab 200 mg IV at Weeks I-0, I-4 and I-8 | IS-2: Period 2: Guselkumab 200 mg IV at Weeks I-12, I-16 and I-20 | IS-2: Period 2: Guselkumab 200 mg SC at Weeks I-12, I-16 and I-20 | MS: Randomized: Placebo SC Every 4 Weeks (q4w) | MS: Randomized: Guselkumab 100 mg SC q8w | MS: Randomized: Guselkumab 200 mg SC q4w | MS: Nonrandomized: Placebo SC q4w | MS: Nonrandomized: Guselkumab 200 mg SC q4w | MS: Dose Adjustment: Placebo SC q4w to Guselkumab 200 mg SC q4w | MS: Dose Adjustment: Guselkumab 100 mg SC q8w to Guselkumab 200 mg SC q4w | MS: Dose Adjustment: Guselkumab 200 mg SC q4w to Guselkumab 200 mg SC q4w
All-Cause Mortality (participants affected / at risk) | 0/109 | 0/108 | 0/111 | 0/67 | 0/79 | 2/296 | 1/440 | 0/172 | 0/129 | 0/203 | 0/197 | 0/199 | 0/122 | 0/125 | 0/75 | 0/23 | 0/31
Serious Adverse Events (participants affected / at risk) | 7/108 | 1/108 | 3/111 | 2/67 | 3/79 | 21/295 | 13/440 | 4/171 | 3/129 | 3/203 | 5/197 | 12/199 | 13/122 | 7/125 | 2/75 | 1/23 | 2/31
Other Adverse Events (participants affected / at risk) | 49/108 | 33/108 | 38/111 | 17/67 | 15/79 | 88/295 | 118/440 | 38/171 | 37/129 | 112/203 | 93/197 | 109/199 | 69/122 | 76/125 | 28/75 | 14/23 | 20/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IS-1: Period 1: Placebo IV at Weeks I-0, I-4 and I-8 (N=108) | IS-1: Period 1: Guselkumab 200 mg IV at Weeks I-0, I-4 and I-8 (N=108) | IS-1: Period 1: Guselkumab 400 mg IV at Weeks I-0, I-4 and I-8 (N=111) | IS-1: Period 2: Guselkumab 200 mg IV at Weeks I-12, I-16 and I-20 (N=67) | IS-1: Period 2: Guselkumab 200 mg SC at Weeks I-12, I-16 and I-20 (N=79) | IS-2: Period 1: Placebo IV at Weeks I-0, I-4 and I-8 (N=295) | IS-2: Period 1: Guselkumab 200 mg IV at Weeks I-0, I-4 and I-8 (N=440) | IS-2: Period 2: Guselkumab 200 mg IV at Weeks I-12, I-16 and I-20 (N=171) | IS-2: Period 2: Guselkumab 200 mg SC at Weeks I-12, I-16 and I-20 (N=129) | MS: Randomized: Placebo SC Every 4 Weeks (q4w) (N=203) | MS: Randomized: Guselkumab 100 mg SC q8w (N=197) | MS: Randomized: Guselkumab 200 mg SC q4w (N=199) | MS: Nonrandomized: Placebo SC q4w (N=122) | MS: Nonrandomized: Guselkumab 200 mg SC q4w (N=125) | MS: Dose Adjustment: Placebo SC q4w to Guselkumab 200 mg SC q4w (N=75) | MS: Dose Adjustment: Guselkumab 100 mg SC q8w to Guselkumab 200 mg SC q4w (N=23) | MS: Dose Adjustment: Guselkumab 200 mg SC q4w to Guselkumab 200 mg SC q4w (N=31)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute Abdomen (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal Fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis Ulcerative (Gastrointestinal disorders) | 4 | 0 | 1 | 1 | 2 | 15 | 6 | 1 | 1 | 1 | 1 | 1 | 2 | 2 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea Haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inflammatory Bowel Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intestinal Perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal Prolapse Syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pancreatitis Chronic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Umbilical Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis Chronic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Adenovirus Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anal Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bacterial Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Clostridium Difficile Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Complicated Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cytomegalovirus Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes Zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic Inflammatory Disease (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rotavirus Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Craniocerebral Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Incarcerated Incisional Hernia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Incisional Hernia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Postoperative Respiratory Failure (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Clear Cell Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fibroadenoma of Breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Guillain-Barre Syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhagic Stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Transient Ischaemic Attack (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute Psychosis (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Calculus Urinary (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Labia Enlarged (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vaginal Polyp (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertensive Emergency (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IS-1: Period 1: Placebo IV at Weeks I-0, I-4 and I-8 (N=108) | IS-1: Period 1: Guselkumab 200 mg IV at Weeks I-0, I-4 and I-8 (N=108) | IS-1: Period 1: Guselkumab 400 mg IV at Weeks I-0, I-4 and I-8 (N=111) | IS-1: Period 2: Guselkumab 200 mg IV at Weeks I-12, I-16 and I-20 (N=67) | IS-1: Period 2: Guselkumab 200 mg SC at Weeks I-12, I-16 and I-20 (N=79) | IS-2: Period 1: Placebo IV at Weeks I-0, I-4 and I-8 (N=295) | IS-2: Period 1: Guselkumab 200 mg IV at Weeks I-0, I-4 and I-8 (N=440) | IS-2: Period 2: Guselkumab 200 mg IV at Weeks I-12, I-16 and I-20 (N=171) | IS-2: Period 2: Guselkumab 200 mg SC at Weeks I-12, I-16 and I-20 (N=129) | MS: Randomized: Placebo SC Every 4 Weeks (q4w) (N=203) | MS: Randomized: Guselkumab 100 mg SC q8w (N=197) | MS: Randomized: Guselkumab 200 mg SC q4w (N=199) | MS: Nonrandomized: Placebo SC q4w (N=122) | MS: Nonrandomized: Guselkumab 200 mg SC q4w (N=125) | MS: Dose Adjustment: Placebo SC q4w to Guselkumab 200 mg SC q4w (N=75) | MS: Dose Adjustment: Guselkumab 100 mg SC q8w to Guselkumab 200 mg SC q4w (N=23) | MS: Dose Adjustment: Guselkumab 200 mg SC q4w to Guselkumab 200 mg SC q4w (N=31)
Anaemia (Blood and lymphatic system disorders) | 11 | 8 | 9 | 4 | 2 | 20 | 22 | 4 | 6 | 5 | 5 | 6 | 5 | 6 | 3 | 2 | 0
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 3 | 0 | 0 | 2 | 0 | 2 | 4 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 5 | 1 | 2 | 0 | 0 | 5 | 2 | 0 | 2 | 2 | 5 | 1 | 1 | 0 | 0 | 0 | 0
Motion Sickness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 3 | 4 | 3 | 1 | 0 | 6 | 4 | 1 | 2 | 4 | 5 | 6 | 1 | 3 | 1 | 1 | 1
Colitis Ulcerative (Gastrointestinal disorders) | 3 | 1 | 3 | 2 | 3 | 12 | 5 | 7 | 7 | 59 | 20 | 26 | 26 | 21 | 7 | 2 | 5
Colon Dysplasia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 4 | 1 | 0 | 0 | 1 | 3 | 0 | 0 | 3 | 3 | 2 | 2 | 2 | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 1 | 1 | 1 | 3 | 2 | 1 | 0 | 1 | 1 | 1 | 3 | 3 | 1 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0 | 1 | 4 | 1 | 1 | 1 | 1 | 0 | 3 | 2 | 0 | 2 | 1
Haemorrhoids Thrombosed (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 5 | 1 | 0 | 0 | 1 | 3 | 2 | 1 | 0 | 6 | 1 | 2 | 2 | 2 | 0 | 0 | 0
Injection Site Erythema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 4 | 0 | 2 | 1 | 0 | 1
Injection Site Hypersensitivity (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Injection Site Induration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection Site Reaction (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 2 | 0 | 0 | 0
Pyrexia (General disorders) | 5 | 2 | 1 | 1 | 2 | 3 | 8 | 1 | 1 | 6 | 7 | 9 | 4 | 8 | 1 | 1 | 1
Hepatic Function Abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Acute Sinusitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Candida Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Covid-19 (Infections and infestations) | 5 | 6 | 2 | 1 | 1 | 13 | 22 | 13 | 9 | 28 | 28 | 20 | 19 | 23 | 5 | 3 | 2
Herpes Virus Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 4 | 1 | 0 | 2 | 2 | 2 | 2 | 6 | 0 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 0 | 1 | 0 | 0 | 8 | 6 | 5 | 3 | 10 | 8 | 7 | 9 | 7 | 3 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 1 | 0 | 1 | 2 | 3 | 0 | 4 | 2 | 0 | 0
Tinea Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 3 | 2 | 0 | 5 | 0 | 2 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 1 | 3 | 0 | 1 | 5 | 2 | 1 | 8 | 6 | 15 | 2 | 5 | 2 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 1 | 7 | 0 | 1 | 2 | 2 | 4 | 3 | 1 | 0 | 1 | 0
Viral Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 1 | 1 | 0
White Blood Cell Count Increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Iron Deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 2 | 2 | 2 | 0 | 3 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 4 | 1 | 1 | 6 | 7 | 2 | 2 | 13 | 12 | 16 | 5 | 5 | 1 | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 8 | 2 | 5 | 3 | 0 | 1 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 0 | 0 | 2 | 4 | 0 | 2 | 0 | 2 | 3 | 1 | 3 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 8 | 3 | 6 | 2 | 3 | 8 | 13 | 1 | 0 | 12 | 8 | 9 | 8 | 5 | 3 | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 1 | 1
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Ejaculation Disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 1 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 1
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 3 | 1 | 0 | 0 | 4 | 9 | 2 | 1 | 2 | 3 | 4 | 4 | 2 | 1 | 0 | 0
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2022-09-12): https://cdn.clinicaltrials.gov/large-docs/45/NCT04033445/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-08): https://cdn.clinicaltrials.gov/large-docs/45/NCT04033445/SAP_001.pdf